CLINICAL TRIAL: NCT02895282
Title: Chronobiology and Childhood Obesity in a Mediterranean Spanish Population (ONTIME-JR: Obesity, Nutrigenomics, Timing, Mediterranean, Junior)
Brief Title: Chronobiology and Childhood Obesity in a Mediterranean Spanish Population
Acronym: ONTIME-JR
Status: Completed | Type: Observational
Sponsor: Universidad de Murcia (Other)
Responsible Party: Principal Investigator, PROF. MARTA GARAULET AZA, Full professor of University of Murcia, Universidad de Murcia
Other Study IDs: SAF2014-52480-R
Record Dates: First submitted 2016-06-30; First posted 2016-09-09 (Estimated); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Obesity; Chronobiology Disorders
Keywords: Obesity; Chronobiology; Circadian
MeSH Terms: conditions — Obesity; Chronobiology Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — saliva
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The main objective is to investigate chronobiological aspects of childhood obesity studying the potential relationship between meal patterns and circadian rhythmicity in a cross-sectional sample of obese, overweight and normal weight children/adolescent.

DETAILED DESCRIPTION:
Childhood obesity has more than doubled in children and tripled in adolescents in the past 30 y. As consequence, increasingly children and adolescents suffer from elevated blood pressure, impaired glucose tolerance, hyperinsulinemia, dyslipidemia. Obesity has a multifactorial etiology since there are potentially numerous contributors to its development and progression. Chronobiology, the science that studies periodic (cyclic) changes in living organisms, has been recently proposed as a new and promising topic to investigate. Alterations of circadian (24 h oscillations) system may contribute to obesity and its complications development such as high blood pressure, insulin resistance, altered fasting lipid profile. Conversely, in a vicious manner, obesity has been regarded as a fault in the circadian system explainable by the association with imbalances and fluctuations of hormones/genes expressions rhythms under the influence of body weight changes.

Thus, the study will examine changes in circadian rhythmicity over a week period. The primary end point will be to evaluate differences between obese/overweight and non-obese children in chronotypes and the responses of these parameters to meal patterns. In particular, non-invasive measures that are well-established determinants of chronotypes will form the core endpoints for the study. Well designed and age-appropriate questionnaires will provide further information in order to study correlations with eating, sleeping and sedentary/active behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Age: 8-12 years of age
* Children from schools in the region of Murcia (Spain) who enter voluntarily

Exclusion Criteria:

* Children who take melatonin or sleep drugs

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children from schools who enter voluntarily in Spanish city of Murcia, located on the Southeast coast of the Mediterranean Sea.
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2014-10; Primary Completion 2018-10 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
BMI | At baseline
  A key index for relating weight to height. BMI is a person's weight in kilograms (kg) divided by his or her height in meters squared.

SECONDARY OUTCOMES:
Individual chronotype with the Munich ChronoType Questionnaire | At baseline
  To assess chronotype with a questionnaire that establishes an algorithm which optimises chronotype assessment by incorporating the information on timing of sleep and wakefulness for both work and free days. The timing and duration of sleep are generally independent. However, when the two are analysed separately for work and free days, sleep duration strongly depends on chronotype. In addition, chronotype is both age- and sex-dependent.
Wrist temperature rhythm | At baseline
  Wrist temperature wireless recording is considered a reliable procedure to evaluate circadian rhythmicity, and an index to establish and follow the effects of chronotherapy in normal living subjects.
Rest-activity rhythm | At baseline
  Rest-activity rhythm as assessed using a acceleration data logger UA-004-64 (Onset Computer, Bourne, MA, USA) placed on the non-dominant arm by means of a sports band, with its x axis parallel to the humerus bone. The sensor is programmed to record data every 30 s.
Sleeping characteristics with a 7 days dietary record of night time and day time (siesta) information | At baseline
  24hs record of sleep will be completed during the 7 days of the experiment. Children are instructed to keep a sleep and food diary designed by the University of Murcia Chronobiology Laboratory. The following data will be obtained for every subject on a daily basis: time to bed, time of lights off, nocturnal awakenings lasting more than 10 minutes, sleep offset, the time the participant arose.
Salivary cortisol determinations | At baseline
  Saliva for cortisol measurements is obtained before breakfast (09:00 h), lunch time (14:00 h), and bedtime (23:00 h) the 6th the 7th day of the experimental week using the Salivette system. Cortisol is measured with radioimmunoassay.
Salivary melatonin determinations on weekends the 6th and 7th day of the experimental week | At baseline
  Samples for the measurement of salivary melatonin are obtained before lunch (14:00 h) and at night (1:00 h) the 6th and 7th day of the experimental week.
Food habits with a 7 days dietary record | At baseline
  During the week of the experiment. Data will be obtained for every subject on a daily basis and they will record the variety of foods that they eat with the portion size.
Total energy intake | At baseline
  During the week of the experiment with a software designed for this purpose.
Macronutrient distribution | At baseline
  from the 7 days dietary record, with a software designed for this purpose.
Food variety | At baseline
  from the 7 days dietary record, with a software designed for this purpose.
Glycemic Index | At baseline
  from the 7 days dietary record, with a software designed for this purpose.
Physical activity | Through study completion
  from the 7 days dietary record, with a software designed for this purpose.
Mediterranean Diet Score | At baseline
  From the 7 days dietary record, with a software designed for this purpose.
Food timing with a 7 days dietary record | At baseline
  Children will be instructed to keep a food diary. Data will be obtained for every subject on a daily basis and they will record the time of the three main meals (breakfast, lunch, and dinner).
Light determination | At baseline
  During the week of the experiment with a light detector device in the neck of the children.
DNA collection in saliva | At baseline
  Saliva will be collected to further extraction of DNA the 7th day of the experimental week.
Saliva collection for microflora determinations | At baseline
  Saliva Collection Method is the SalivaBio Oral Swab the 7th day of the experimental week.

CONTACTS AND LOCATIONS:
Overall Officials: Marta Garaulet, PhD, Principal Investigator — University of Murcia. Spain
Locations (2):
- Spain (2):
  - Chronobiology laboratory, Department of Physiology, Murcia
  - University of Murcia, Murcia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Qian J, Martinez-Lozano N, Tvarijonaviciute A, Rios R, Scheer FAJL, Garaulet M. Blunted rest-activity rhythms link to higher body mass index and inflammatory markers in children. Sleep. 2021 May 14;44(5):zsaa256. doi: 10.1093/sleep/zsaa256. PMID 33249510
- [Derived] Barraco GM, Martinez-Lozano N, Vales-Villamarin C, Del Carmen Blaya M, Rios R, Madrid JA, Fardy P, Garaulet M. Circadian health differs between boys and girls as assessed by non-invasive tools in school-aged children. Clin Nutr. 2019 Apr;38(2):774-781. doi: 10.1016/j.clnu.2018.03.001. Epub 2018 Mar 21. PMID 29609867